CLINICAL TRIAL: NCT06821009
Title: Effectiveness of a Cloud-based Digital Health Navigation Program for Colorectal Cancer Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Digital Health Navigation Solutions, Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, David P. Miller, Jr., CEO, Digital Health Navigation Solutions, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IRB00118236; 4R42CA275665 (NIH)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mPATH-CRC (Experimental): Participants randomized to the mPATH arm will receive a text message inviting them to use the mPATH-CRC WebApp. The WebApp verifies individuals are due for routine colorectal cancer (CRC) screening, educates them about their options, and lets them request a screening test via the program.
  Interventions: Other: mPATH-CRC
- Usual Care (Control) (Placebo Comparator): Patients randomized to the control arm will receive usual care, which includes the organizations' standard procedures for addressing CRC screening.
  Interventions: Other: Usual Care (Control)

INTERVENTIONS:
Other: mPATH-CRC — Individuals will receive an automated text message inviting them to use the mPATH-CRC WebApp. The WebApp takes approximately 5 to 8 minutes to complete. The WebApp verifies patients are due for routine CRC screening, educates them about their options, and lets them request a screening test via the program.
  Arms: mPATH-CRC
Other: Usual Care (Control) — Patients randomized to the control arm will receive usual care, which includes the organizations' standard procedures for addressing CRC screening. In the participating Fee-for-Service and Value-Based settings, the EHR flags patients who are overdue for CRC screening as a "care gap" that is visible to all primary care providers.
  Arms: Usual Care (Control)

SUMMARY:
mPATH-CRC (mobile Patient Technology for Health) is an automated direct-to-patient digital health program about colorectal cancer screening. The goal of this project is to test a cloud-based version of mPATH that patients can use at home independent of a scheduled medical visit. Patients will access mPATH on their own devices using a hyperlink sent via text message. The cloud version of mPATH will have the proven effective content of the tablet version, including the ability to request a screening test directly via the program. mPATH will then share this information with the patient's healthcare organization so screening can be arranged. This cloud-based version will be highly scalable, have broad reach, and be easy to support, making it a commercially viable product. This project will (1) test the reach and effectiveness of the mPATH web app in two different healthcare settings: a Fee-for-Service setting, and a value-based care setting; and (2) determine the value generated by mPATH in each healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-74 years
2. Be identified in the electronic health record as due for routine CRC screening, defined as

   1. No colonoscopy in prior 10 years
   2. No flexible sigmoidoscopy in prior 5 years
   3. No CT colography in prior 5 years
   4. No FIT-DNA test (Cologuard) within prior 3 years
   5. No Fecal Occult Blood Test within prior 1 year
3. Have a cell phone number listed in the EHR
4. Have a preferred language of English or Spanish in the EHR
5. Upcoming appointment within 9 to 16 days
6. Georgia Market Only: Insurance type is listed as Medicare Advantage.

Exclusion Criteria

1. Prior diagnosis of colorectal cancer
2. Prior history of total colectomy
3. Currently enrolled in palliative care or Hospice
4. Age over 65 AND currently enrolled in an Institutional SNP (I-SNP) or living in Long Term Care
5. Age over 65 with frailty and advanced illness (as defined by the health system's My Panel metric which mirrors the HEDIS COL-E quality metric for CRC screening)

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6500 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of mPATH-CRC | 180 Days
  The proportion of individuals who complete a CRC screening test (colonoscopy, FIT, or FIT-DNA) within 180 days of randomization in both arms

SECONDARY OUTCOMES:
Reach of mPATH-CRC | 30 Days
  The proportion of patients in the mPATH-CRC arm who complete the mPATH-CRC Web App to the point of being told if screening is due or not due
Reporting current CRC screening | 30 Days
  The proportion of participants within the mPATH arm who report they are current with CRC screening within the mPATH program.
CRC screening ordered | 180 Days
  The proportion of patients who have a CRC screening test ordered within 180 days of randomization in both arms.
Colorectal Neoplasia | 180 days
  The proportion of patients in each arm with neoplasia found on colonoscopy within 180 days after randomization.
Mean revenue generated in a Fee-for-Service setting | 365 Days
  Mean revenue generated in a Fee-for-Service setting from screening and resulting downstream care within 12 months (365 days) of the screening event, assuming Medicare reimbursement rates in both arms.
Quality gaps closed in a value-based care setting | 180 Days
  Proportion of quality gaps closed in a value-based setting in each arm defined as completing screening or acquiring documentation of previously completed screening in both arms.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atrium Health Floyd, Rome, Georgia
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data that underlie our published or presented results.
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of the publication of the study's results. Data will be kept available until 4 years after the publication of the study's results.
Access Criteria: Researchers must provide the investigative team a methodologically sound proposal. Use of the data will be limited to achieve the aims in their submitted proposal. To gain access, data requestors will need to sign a data access agreement.